CLINICAL TRIAL: NCT00306618
Title: A Single-Center, Open-Label, Phase II, Safety, Pharmacokinetic and Efficacy of Panzem Nanocrystal Colloidal Dispersion Administered Orally to Patients With Recurrent Glioblastoma Multiforme
Brief Title: Safety and Efficacy Study of Panzem NCD to Treat Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Chief Medical Officer, EntreMed, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-CLN-005
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2008-12-10 (Estimated); Status verified 2008-12

CONDITIONS: Recurrent Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — 2-Methoxyestradiol

INTERVENTIONS:
Drug: Panzem Nanocrystal Colloidal Dispersion — Panzem NCD suspension, 100 mg/mL, four times daily continuous dosing
  Other Names: 2-methoxyestradiol; 2ME2

SUMMARY:
This single-center, open-label, phase 2 study will evaluate the anti-tumor activity, as well as the safety and pharmacokinetics, of Panzem (2-methoxyestradiol, 2ME2) Nanocrystal Colloidal Dispersion (NCD) administered in patients with recurrent glioblastoma multiforme (GBM)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a 1st or 2nd recurrent/progressive primary WHO grade IV malignant glioma (glioblastoma multiforme or gliosarcoma).
* 18 years or older
* An interval of at least 2 weeks between prior surgical resection or any major surgery or 4 weeks between prior radiotherapy or chemotherapy (except nitrosoureas which require 6 weeks)
* Karnofsky performance score equal to or greater than 70%
* Hematocrit greater than 29%, absolute neutrophil count greater than 1,500 cells/micro liters, platelets greater than 100,000 cells/ micro liters
* Serum creatinine less than 1.5 X upper limit of normal (ULN), serum SGOT less than 2.5 X ULN; and bilirubin less than 1.5 times ULN
* Signed informed consent form and authorization for use and disclosure of protected health information approved by the IRB prior to patient entry
* Agree to use effective contraceptive methods

Exclusion Criteria:

* Current, active systemic bleeding or excessive risk of bleeding
* Be pregnant or lactating; not employing effective birth control
* Concurrent severe and/or uncontrolled medical disease
* Impairment of gastrointestinal (GI) function/disease
* Requirement for therapy with coumadin (warfarin sodium)
* Patient is less than 5 years free of another primary malignancy
* Patients unwilling to or unable to comply with the protocol
* Grade 2 or greater peripheral sensory neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
6 month progression free survival and median overall survival | time of progression; survival

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, M.D., Principal Investigator — The Brain Center at Duke, Duke University Medical Center
Locations (1):
- The Brain Tumor Center, Duke University Medical Center, Durham, North Carolina, United States